CLINICAL TRIAL: NCT03012165
Title: A Study of ADX-102 in Subjects With Allergic Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-102-AC-004
Record Dates: First submitted 2016-12-14; First posted 2017-01-06 (Estimated); Results first posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Conjunctivitis, Allergic
Keywords: ADX-102; Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ADX-102 Ophthalmic Drops (0.5%) (Experimental): ADX-102 Ophthalmic Drops (0.5%) administered twice in two weeks.
  Interventions: Drug: ADX-102 Ophthalmic Drops (0.5%)
- ADX-102 Ophthalmic Drops (0.1%) (Experimental): ADX-102 Ophthalmic Drops (0.1%) administered twice in two weeks.
  Interventions: Drug: ADX-102 Ophthalmic Drops (0.1%)
- Vehicle of ADX-102 Ophthalmic Drops (Placebo Comparator): Vehicle of ADX-102 Ophthalmic Drops
  Interventions: Drug: Vehicle of ADX-102 Ophthalmic Drops

INTERVENTIONS:
Drug: ADX-102 Ophthalmic Drops (0.5%) — ADX-102 Ophthalmic Drops (0.5%) administered twice in two weeks.
  Arms: ADX-102 Ophthalmic Drops (0.5%)
Drug: ADX-102 Ophthalmic Drops (0.1%) — ADX-102 Ophthalmic Drops (0.1%) administered twice in two weeks.
  Arms: ADX-102 Ophthalmic Drops (0.1%)
Drug: Vehicle of ADX-102 Ophthalmic Drops — Vehicle of ADX-102 Ophthalmic Drops administered twice in two weeks.
  Arms: Vehicle of ADX-102 Ophthalmic Drops

SUMMARY:
A Multi-Center, Double-Masked, Randomized, Vehicle-Controlled, Phase 2b Evaluation of the Onset and Duration of ADX-102 Ophthalmic Drops (0.5% and 0.1%) Compared to Vehicle of ADX-102 Ophthalmic Drops in the Conjunctival Allergen Challenge (Ora-CAC®) Model of Acute Allergic Conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age of either gender and any race
* have a positive history of ocular allergies and a positive skin test reaction to a seasonal (grasses, ragweed, and/or trees) or perennial allergen (cat dander, dog dander, dust mites, cockroach) as confirmed by an allergic skin test within the past 24 months
* have a calculated visual acuity of 0.7 logMAR or better in each eye as measured using an ETDRS chart

Exclusion Criteria:

* have known contraindications or sensitivities to the use of the investigational product or any of its components
* have any ocular condition that, in the opinion of the investigator, could affect the subject's safety or trial parameters (including but not limited to narrow angle glaucoma, clinically significant blepharitis, follicular conjunctivitis, iritis, pterygium or a diagnosis of dry eye)
* have had ocular surgical intervention within three (3) months prior to Visit 1 or during the study and/or a history of refractive surgery within the past six (6) months
* have a known history of retinal detachment, diabetic retinopathy, or active retinal disease
* have the presence of an active ocular infection (bacterial, viral or fungal) or positive history of an ocular herpetic infection at any visit
* be a female who is currently pregnant, planning a pregnancy, lactating, not using a medically acceptable form of birth control throughout the study duration and for 14 days prior to the installation of investigational product, or has a positive urine pregnancy test at Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-12; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Eye Care Centers Management, Morrow, Georgia
  - Silverstein Eye Centers, Kansas City, Missouri
  - Apex Eye Clinical Research, Mason, Ohio
  - Philadelphia Eye Associates, Philadelphia, Pennsylvania
  - Total Eye Care, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ADX-102 Ophthalmic Drops (0.5%) | ADX-102 Ophthalmic Drops (0.1%) | Vehicle of ADX-102 Ophthalmic Drops
Started | 53 | 51 | 50
Completed | 51 | 49 | 49
Not Completed | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ADX-102 Ophthalmic Drops (0.5%) | ADX-102 Ophthalmic Drops (0.1%) | Vehicle of ADX-102 Ophthalmic Drops | Total
Number analyzed (Participants) | 53 | 51 | 50 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 51 | 47 | 48 | 146
  >=65 years | 2 | 4 | 2 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 27 | 30 | 97
  Male | 13 | 24 | 20 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 3 | 12
  Not Hispanic or Latino | 49 | 46 | 46 | 141
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 34 | 34
  Black or African American | 18 | 17 | 13 | 48
  White | 35 | 33 | 0 | 68
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 2
Iris Color (Right Eye) [Number; unit: participants]
  Black | 0 | 0 | 1 | 1
  Blue | 8 | 11 | 10 | 29
  Brown | 31 | 29 | 26 | 86
  Hazel | 6 | 5 | 7 | 18
  Green | 8 | 5 | 6 | 19
  Gray | 0 | 1 | 0 | 1
  Other | 0 | 0 | 0 | 0
Iris Color (Left Eye) [Number; unit: participants]
  Black | 0 | 0 | 1 | 1
  Blue | 8 | 11 | 10 | 29
  Brown | 31 | 29 | 26 | 86
  Hazel | 6 | 5 | 7 | 18
  Green | 8 | 5 | 6 | 19
  Gray | 0 | 1 | 0 | 1
  Other | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching Evaluated by the Subject at 10(±1) Minutes Post the Ora Calibra® Conjunctival Allergen Challenge at Day 15.
Description: Ocular itching using the Ora Calibra® Conjunctival Allergen Challenge Ocular Itching Scale (0 = least, 4= most), where a higher score is indicative of a worse outcome. The intervention was administered bilaterally.
Time Frame: Efficacy assessment period (Day 1 through Day 15), Day 15 reported.
Population: Intent to treat population with observed data only.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ADX-102 (0.5%): ADX-102 Ophthalmic Drops (0.5%) administered twice in two weeks.
  ADX-102 Ophthalmic Drops (0.5%): ADX-102 Ophthalmic Drops (0.5%) administered twice in two weeks.
- ADX-102 (0.1%): ADX-102 Ophthalmic Drops (0.1%) administered twice in two weeks.
  ADX-102 Ophthalmic Drops (0.1%): ADX-102 Ophthalmic Drops (0.1%) administered twice in two weeks.
- Vehicle: Vehicle of ADX-102 Ophthalmic Drops
  Vehicle of ADX-102 Ophthalmic Drops: Vehicle of ADX-102 Ophthalmic Drops administered twice in two weeks.
Arm/Group | ADX-102 (0.5%) | ADX-102 (0.1%) | Vehicle
Number analyzed (Participants) | 51 | 49 | 49
units on a scale | 2.020 (0.9821) | 2.398 (0.8290) | 2.515 (0.9661)

2. Primary Outcome: Ocular Itching Evaluated by the Subject at 15(±1) Minutes Post the Ora Calibra® Conjunctival Allergen Challenge at Day 15.
Description: as for outcome 1
Time Frame: Efficacy assessment period (Day 1 through Day 15), Day 15 reported.
Population: Intent to treat population with observed data only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADX-102 (0.5%) | ADX-102 (0.1%) | Vehicle
Number analyzed (Participants) | 51 | 49 | 49
units on a scale | 1.662 (1.0085) | 1.801 (0.9601) | 1.985 (0.9768)

3. Primary Outcome: Ocular Itching Evaluated by the Subject at 20(±1) Minutes Post the Ora Calibra® Conjunctival Allergen Challenge at Day 15.
Description: as for outcome 1
Time Frame: Efficacy assessment period (Day 1 through Day 15), Day 15 reported.
Population: Intent to treat with observed data only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADX-102 (0.5%) | ADX-102 (0.1%) | Vehicle
Number analyzed (Participants) | 51 | 49 | 49
units on a scale | 1.152 (0.9799) | 1.434 (0.9773) | 1.551 (1.0433)

ADVERSE EVENTS:
Time Frame: Adverse event data was captured for approximately 5 weeks for each subject during clinical trial participation.
Arm/Group | ADX-102 Ophthalmic Drops (0.5%) | ADX-102 Ophthalmic Drops (0.1%) | Vehicle of ADX-102 Ophthalmic Drops
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/51 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/51 | 0/49
Other Adverse Events (participants affected / at risk) | 0/53 | 0/51 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT03012165/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT03012165/SAP_001.pdf